CLINICAL TRIAL: NCT03144973
Title: Meaning of Periodontitis in Post-operative Complications After Upper Gastrointestinal Tract Surgery
Brief Title: Periodontitis and Upper gi Post-operative Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Tiina Vuorela, MD, PHD student, Junior surgeon, Helsinki University Central Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: HUS/269/2017
Record Dates: First submitted 2017-05-03; First posted 2017-05-09 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Periodontitis; Surgery--Complications
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: All the patients that have upper-gi surgery in our time frame are asked to join in the study
Who Masked: Care Provider
Masking Description: operating surgeons or surgeons in the surgical ward do not get to know the test result so it won't affect in patient care
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: periosafe — mouth rinsing quick-test

SUMMARY:
Periodontitis is a infection of mouth gingival mucosa and connecting tissue. It has been shown in previous studies to have a effect on the risk of heart diseases getting worse and elevate risk in heart surgery. The investigators are studying periodontitis and how it affects upper gastrointestinal tract patients complication rates and the quality of complications.

DETAILED DESCRIPTION:
Before patricipating patients go to preop, the investigators have them take a mouth rinsing quick-test, periosafe(c), that tells specifically about periodontitis. Participants go to surgery (upper gi) and have a normal operation following our clinics standards and normal follow up. After the investigators analyze the patient data concerning possible complications and do they have relations between the positive periodontitis results. Participants are also given advice about seeing a dentist if positive results are seen, but the operating surgeons do not get to know the mouth rinsing test results.

ELIGIBILITY:
Inclusion Criteria:

* Need for a upper gi surgery

Exclusion Criteria:

-

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
meaning of periodontitis in post operative complications | 1 month after surgery
  Periodontitis is being tested by Periosafe (c) quick-test. Participants with positive results on the test have periodontitis. Participants patient data is being analyzed after surgery and is compared to periodontitis results. The correlation between periodontitis and surgical complications is subject to analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Seppänen, Phd, Dos, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki university hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No